CLINICAL TRIAL: NCT06007391
Title: Pilot Study of Tolerance and Efficacy Nicotinamide (vitamin B3) in Dominant Optic Atrophy OPA1
Brief Title: Tolerance and Efficacy Nicotinamide (vitamin B3) in Dominant Optic Atrophy OPA1
Acronym: NICOPA1-TOL
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49RC23_0195
Record Dates: First submitted 2023-07-06; First posted 2023-08-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Nicotinamide Adverse Reaction
MeSH Terms: interventions — Niacinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- nicotinamide (Experimental)
  Interventions: Drug: Nicotinamide

INTERVENTIONS:
Drug: Nicotinamide — nicotinamide 3g per day

SUMMARY:
Dominant Optic Atrophy (hereafter known as DOA) is a neurodegenerative pathology of the optic nerve inducing progressive loss of central visual field and visual acuity. There is currently no proven treatment for this disease. The metabolomics work of Pascal Reynier's team revealed a specific metabolomic signature of DOA in the plasma of patients. This metabolomic signature revealed a relative deficiency in nicotinamide compared to a control population, a vitamin compound (vitamin B3) known to be neuroprotective for the optic nerve and mitochondria. Note that the investigator have also identified this nicotinamide deficiency in primary open-angle glaucoma and Leber's hereditary optic neuropathy, the other most common cause of hereditary optic neuropathy, these three optic nerve conditions sharing a common pathophysiological mechanism of mitochondrial deficit. In addition, an American team demonstrated the high neuroprotective power on the optic nerve of nicotinamide in a mouse model of glaucoma. These arguments converge towards the potential therapeutic interest of this vitamin in degenerative pathologies of the optic nerve. This is encouraged by the fact that two randomized clinical trials have confirmed a benefit of nicotinamide in glaucoma. The objective of this pilot study is to test the tolerance and efficacy of nicotinamide in DOA and DOA+ patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients with DOA or DOA+ due to a heterozygous pathogenic variant in the OPA1 gene
* Naïve patients (> 3 months) in terms of taking nicotinamide
* Patients able to take oral medication and comply with specific study procedures
* Patients affiliated or beneficiaries of a social security scheme
* Signature of voluntary, free and informed consent to participate in the study

Exclusion Criteria:

* Asymptomatic patients (= healthy carriers of an OPA1 mutation but not having developed optic neuropathy)
* Patients with another associated severe ophthalmological pathology (advanced glaucoma, retinal pathology, etc.)
* Patients treated with Idebenone
* Patients with a level of transaminase(s) (ASAT and/or ALAT) twice higher than the high normal value.
* Pregnant, breastfeeding or parturient women
* Patients with a contraindication to nicotinamide
* Persons deprived of liberty by administrative or judicial decision
* Patients subject to a legal protection measure
* Persons undergoing psychiatric treatment under duress
* Persons unable to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of patient with neurologic or ophtalmological adverse event | at 6 months
  photopic negative response PhNR, optical coherence tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No